CLINICAL TRIAL: NCT06586671
Title: An Open-Label, Two-Part, Two-Period Crossover Study to Determine Bioequivalence Between Nemtabrutinib FFP and FMF2 Formulations & FMF1 and FMF2 Formulations at 65 mg Single Dose in Healthy Male Participants
Brief Title: A Study to Compare Forms of Nemtabrutinib (MK-1026) in Healthy Adult Participants (MK-1026-007)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1026-007; MK-1026-007 (Other: MSD)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — ARQ531

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nemtabrutinib Form A (Experimental): Participants receive nemtabrutinib form A orally.
  Interventions: Drug: Nemtabrutinib
- Nemtabrutinib Form B (Experimental): Participants receive nemtabrutinib form B orally.
  Interventions: Drug: Nemtabrutinib
- Nemtabrutinib Form C (Experimental): Participants receive nemtabrutinib form C orally.
  Interventions: Drug: Nemtabrutinib

INTERVENTIONS:
Drug: Nemtabrutinib — Oral administration
  Other Names: MK-1026; ARQ-531

SUMMARY:
The goal of the study is to measure and compare the levels of nemtabrutinib in the blood after taking different forms of nemtabrutinib orally on an empty stomach (fasted) to see if they are the same or different.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body mass index (BMI) ≥18 and ≤32 kg/m^2, inclusive

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer with pre-specified exceptions (adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix or other malignancies that have been successfully treated with appropriate follow up and therefore unlikely to recur for the duration of the study, per protocol guidelines)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Parts 1 and 2: Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Nemtabrutinib | At designated time points (up to approximately 2 weeks)
  Blood samples will be collected to determine the AUC0-inf of nemtabrutinib.
Parts 1 and 2: Maximum Plasma Concentration (Cmax) of Nemtabrutinib | At designated time points (up to approximately 2 weeks)
  Blood samples will be collected to determine the Cmax of nemtabrutinib.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 2 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 2 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- QPS-MRA, LLC-Early Phase (Site 0002), South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com